CLINICAL TRIAL: NCT01053442
Title: Absorption, Stable Isotope Appearance and NTBI Profile From NaFeEDTA and Ferrous Sulphate
Brief Title: Absorption, Stable Isotope Appearance and Non-transferrin-bound Iron (NTBI) Profile From NaFeEDTA and Ferrous Sulphate
Acronym: SIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: DSM Nutritional Products, Inc. (Industry)
Responsible Party: Principal Investigator, Prof. Michael B. Zimmermann, Prof, Swiss Federal Institute of Technology
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: ETHZ-SIA2
Record Dates: First submitted 2010-01-20; First posted 2010-01-21 (Estimated); Last update posted 2012-04-05 (Estimated); Status verified 2012-04

CONDITIONS: Iron Deficiency
Keywords: iron absorption; stable isotopes; NaFeEDTA; Non-transferrin-bound iron (NTBI); Hepcidin
MeSH Terms: conditions — Iron Deficiencies

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- NaFeEDTA (Experimental): The maize porridge is fortified with 2.5mg iron as NaFeEDTA
  Interventions: Dietary Supplement: Porridge fortified with either NaFeEDTA
- FeSO4 (Active Comparator): The maize porridge is fortified with 2.5 mg iron as ferrous sulphate plus ascorbic acid.
  Interventions: Dietary Supplement: FeSO4

INTERVENTIONS:
Dietary Supplement: Porridge fortified with either NaFeEDTA — 265g maize porridge is fortified with 2.5 mg iron as NaFeEDTA.
  Arms: NaFeEDTA
Dietary Supplement: FeSO4 — Maize porridge is fortified with 2.5 mg iron as ferrous sulphate and 45 mg ascorbic acid.
  Arms: FeSO4

SUMMARY:
Several iron compounds are used for fortification, including ferrous sulphate and NaFeEDTA. The absorption profile of these may differ because of differences in their dissolution in the gastrointestinal tract and in their interaction with dietary inhibitors of iron absorption. As these differences might lead result in varying reactions in the blood stream, the appearance rate of the stable iron isotope, hepcidin, non-transferrin-bound iron and total iron in the plasma will be monitored over six hours in adult women. This is relevant as a spike of absorbed iron may increase non-transferrin-bound iron and this could be pro-oxidative or increase growth of pathogens. Hepcidin is a key mediator of iron absorption and will help explain the potential differences in the plasma iron profile.

The use of stable iron isotope appearance curves to specifically detect the appearance of small amounts of absorbed iron in the blood and distinguish between circulating body iron and iron absorbed from the test meal was tested in a pilot study (EK 2008-23). This method is now used in a bigger sample to test the differences in absorption profile of ferrous sulphate, FePPi and NaFeEDTA given at fortification level with a meal.

ELIGIBILITY:
Inclusion Criteria:

* Serum ferritin <60 ug/ l, haemoglobin > 100 g/ l
* Women
* < 65 kg body weight
* Healthy

Exclusion Criteria:

* Pregnant or lactating
* Taking iron supplements

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2010-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Stable iron isotope appearance in the plasma over 8 hours | day 1: 0', 30', 60', 120', 240', 480', day 8 0', 30', 60', 120', 240', 480'

SECONDARY OUTCOMES:
Isotope incorporation with erythrocytes | day 22

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratory of Human Nutrition, Zurich, Canton of Zurich, Switzerland